CLINICAL TRIAL: NCT05613465
Title: A Double-blind, Randomized Controlled Study of Adjuvant Chemotherapy Plus Codonopsis Pilosula Nnannf /Placebo After Radical Surgery
Brief Title: Adjuvant Chemotherapy Plus Codonopsis Pilosula Nnannf /Placebo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZJPPHGIP-RCT202210
Record Dates: First submitted 2022-10-31; First posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Pancreatic Carcinoma; Adjuvant Chemotherapy; Cancer-related Fatigue
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): Codonopsis pilosula Nnannf
  Interventions: Drug: Codonopsis
- Control group (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Codonopsis — Codonopsis pilosula Nnannf is oral liquid, which has been approved for listing
  Arms: intervention
Drug: Placebo — Placebo is packaged in the same package as the drug
  Arms: Control group

SUMMARY:
Pancreatic carcinoma patients got benefit from adjuvant therapy after radical surgery. Gemcitabine combined with albumin-paclitaxel was recommended as the first-line regimen for adjuvant chemotherapy by NCCN guidelines. The most common non-hematological adverse events associated with gemcitabine combined with albumin-paclitaxel treatment were fatigue (54%), followed by alopecia (50%), and grade 3 or higher adverse events were mainly granulocytopenia, leukopenia, fatigue, and peripheral nerve damage. Cancer-related fatigue (CRF) is the most common concomitant symptom in cancer patients, especially during chemotherapy, which has a negative impact on patients' work, social relationships, emotions and daily activities. Therefore, it is of great clinical significance to improve CRF in cancer patients. From the perspective of traditional Chinese medicine, CRF patients will have a series of syndromes such as low function of viscera, general weakness, and emaciation, which last for more than 2 weeks and affect patients' physiology and psychology at the same time. Codonopsis pilosula Nnannf can restore the postoperative immune ability of patients as soon as possible after chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pancreatic adenocarcinoma was confirmed by pathology after radical resection.
* Patients received adjuvant chemotherapy after surgery, and the chemotherapy regimen was gemcitabine combined with albumin paclitaxel.
* ECOG score was less than 2.
* The expected survival time was more than 3 months.

Exclusion Criteria:

* Patients were received radiotherapy, chemotherapy within 4 weeks.
* Pregnant and lactating women.
* Patients were known to be allergic to the regimen.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10-25 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Cancer-related fatigue | 9 weeks
  The revised Piper fatigue scale (PFS⁃R) was used for accessing Cancer-related fatigue

SECONDARY OUTCOMES:
Immunologic function | 9 weeks
  Number of T cell subgroups、B cells and NK cells count in plasma were measured every three weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Provincial People'S Hospital, Hangzhou, Other (Non U.s.), China